CLINICAL TRIAL: NCT01052012
Title: Bupivacaine Effectiveness and Safety in SABER Trial (BESST)
Brief Title: Bupivacaine Effectiveness and Safety in SABER® Trial
Acronym: BESST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C803-025
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Abdominal Surgery
Keywords: Postoperative pain; Post-operative pain; Opioid; Laparoscopic surgery; Bupivacaine; Local anesthetic
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active: SABER-Bupivacaine (Experimental): SABER-Bupivacaine
  Interventions: Drug: SABER-Bupivacaine
- Comparator: Bupivacaine HCl (Active Comparator): Bupivacaine HCl
  Interventions: Drug: Bupivacaine HCl
- Placebo: SABER-Placebo (Placebo Comparator): SABER-Placebo
  Interventions: Drug: SABER-Placebo

INTERVENTIONS:
Drug: SABER-Bupivacaine — Injectable Extended Release Solution; SABER-Bupivacaine /Once
  Other Names: POSIMIR® bupivacaine solution
  Arms: Active: SABER-Bupivacaine
Drug: Bupivacaine HCl — Injectable Solution; Bupivacaine HCl /Once
  Arms: Comparator: Bupivacaine HCl
Drug: SABER-Placebo — Injectable Solution; SABER-Placebo/Once
  Arms: Placebo: SABER-Placebo

SUMMARY:
This is a research study testing SABER-Bupivacaine (an experimental pain-relieving medication). SABER-Bupivacaine is designed to continuously deliver bupivacaine, a common local anesthetic, for a few days in order to treat local post-surgical pain.

The purpose of this study is to investigate safety (side effects) associated with the use of SABER-Bupivacaine and how well it works in reducing pain and opioid-related side effects following various kinds of abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to read and understand the consent form, provide written consent, complete trial-related procedures, and communicate with the trial staff
* Males and females, 18 years of age and older scheduled to undergo elective general abdominal surgery
* Patients must be healthy or have only mild systemic disease
* BMI < 45
* Patients must have ECG wave form within normal limits
* Female and male patients must agree to use medically acceptable method of contraception throughout the entire trial period and for 1 week after the trial participation is completed

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients undergoing emergency surgery (unless full consent is obtained and all screening procedures are completed prior to surgery)
* Significant concomitant surgical procedure
* History of multiple prior laparotomy procedures
* Cancer with known metastases pre-operatively, which are suspected to impact post-operative recovery or pain
* Planned formation of stoma during surgery or plans to undergo another laparotomy procedure within 30 days post-operatively
* Pre-operative evidence of sepsis or septic shock
* Pre-operative evaluation that suggests a surgery may preclude full closure of the incision(s)
* Patients with current or regular use of systemic steroids, anticonvulsants, antiepileptics, antidepressants, or monoamine oxidase inhibitors, who cannot be withdrawn from these medications
* Patients with current or regular use of drugs known to significantly prolong the QTc interval
* Patients with known hypersensitivity to local anesthetic agents of the amide type (e.g. lidocaine, bupivacaine)
* Patients with known hypersensitivity to morphine
* Patients with conditions contraindicated for use of opioids
* Patients with atrial fibrillation/flutter or other non-sinus rhythm (including paced rhythm); left bundle branch block (LBBB); or the following conditions: right bundle branch block (RBBB) in presence of a cardiac disease, significant cardiomyopathy, and myocardial infarction within last 6 months
* Patients with a serum creatinine level two times more than the local laboratory normal limit
* Patients who have received greater than 600 mg morphine equivalent daily dose for three or more days per week in the month prior to the surgical procedure
* Patients who are currently being treated with methadone, or history of methadone use within the previous 6 months
* Patients with known or suspected abuse of opioids or other illicit drugs
* Patients with known or suspected alcohol abuse
* Participation in another clinical trial at the same time or within 30 days of this trial
* Patients who, in the Investigator's opinion, should not participate in the trial or may not be capable of following the trial schedule for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Durect
Locations (25):
- United States (21):
  - DURECT Study Site, Birmingham, Alabama
  - DURECT Study Site, Florence, Alabama
  - DURECT Study Site, Mobile, Alabama
  - DURECT Study Site, Montgomery, Alabama
  - DURECT Study Site, Sheffield, Alabama
  - DURECT Study Site, Arcadia, California
  - DURECT Study Site, Fontana, California
  - DURECT Study Site, Laguna Hills, California
  - DURECT Study Site, Pasadena, California
  - DURECT Study Site, Tampa, Florida
  - DURECT Study Site, Powder Springs, Georgia
  - DURECT Study Site, Indianapolis, Indiana
  - DURECT Study Site, Boston, Massachusetts
  - DURECT Study Site, Troy, Michigan
  - DURECT Study Site, Duluth, Minnesota
  - DURECT Study Site, New York, New York
  - DURECT Study Site, Durham, North Carolina
  - DURECT Study Site, Columbus, Ohio
  - DURECT Study Site, Hershey, Pennsylvania
  - DURECT Study Site, Houston, Texas
  - DURECT Study Site, Temple, Texas
- Australia (3):
  - DURECT Study Site, Woodville South, South Australia
  - DURECT Study Site, Box Hill, Victoria
  - DURECT Study Site, Ringwood East, Victoria
- DURECT Study Site, Christchurch, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 15 sites in the US, 3 sites in Australia, and 1 site in New Zealand. The study was initiated on 21 December 2009 and completed on 30 September 2011.
Pre-assignment Details: total of 393 patients were screened and 331 patients were randomized. There were 26 patients who were randomized but not treated. The reasons for not treating these patients included: conditions encountered during surgery necessitated procedures that did not meet protocol requirements, peri-operative epidural analgesia was administered, the test drug was not available, or the patient withdrew consent
Groups:
- Cohort 1-POSIMIR; Cohort 1-Bupivacaine HCl: Open Laparotomy
- Cohort 2-POSIMIR; Cohort 2-Bupivacaine HCl: Laparoscopic Cholecystectomy
- Cohort 3-POSIMIR; Cohort 3-Placebo: Laparoscopic Assisted Colectomy
Period: Overall Study
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Started | 32 | 23 | 30 | 20 | 140 | 86
Completed | 28 | 17 | 30 | 19 | 124 | 76
Not Completed | 4 | 6 | 0 | 1 | 16 | 10
Not completed — Not treated | 2 | 5 | 0 | 0 | 11 | 8
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo | Total
Number analyzed (Participants) | 30 | 18 | 30 | 20 | 129 | 78 | 305
Age, Continuous [Mean (Full Range); unit: years] | 56.8 [28 to 85] | 53.8 [22 to 87] | 44.2 [23 to 74] | 39.5 [24 to 64] | 60.2 [24 to 87] | 58.2 [34 to 84] | 56.1 [22 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 20 | 14 | 70 | 34 | 165
  Male | 12 | 9 | 10 | 6 | 59 | 44 | 140
BMI [Mean (Full Range); unit: kg/m^2] | 30.5 [17.2 to 52.5] | 27.0 [20.2 to 36.1] | 30.8 [20.7 to 42.2] | 31.9 [19.2 to 44.8] | 29.4 [15.9 to 46.8] | 27.5 [14.4 to 37.9] | 29.2 [14.1 to 52.5]

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity on Movement
Description: Mean pain intensity on movement AUC (time-normalized AUC) during the period 0 to 72 hours post-dose. Pain intensity was assessed with a standard 0 to 10 numeric rating scale (NRS), where no pain at all was rated as 0 and the worst pain imaginable was rated as 10. The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 0 to 72 hours post-dose
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
score on a scale | 4.9 [4.0 to 5.7] | 5.0 [4.7 to 6.8] | 2.8 [2.0 to 3.6] | 3.9 [3.0 to 4.8] | 4.8 [4.4 to 5.2] | 5.1 [4.7 to 5.6]
Statistical Analysis 1: Comparison: Cohort 1-POSIMIR vs Cohort 1-Bupivacaine HCl; Test type: Superiority; p = 0.1473, ANCOVA; With pooled site and treatment group as factors and incision length as a covariate; LS Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-2.11 to 0.33], Standard Error of Mean 0.597
Statistical Analysis 2: Comparison: Cohort 2-POSIMIR vs Cohort 2-Bupivacaine HCl; Test type: Superiority; p = 0.0601, ANCOVA; with pooled site and treatment group as factors and incision length as a covariate; LS Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-2.16 to 0.05], Standard Error of Mean 0.547
Statistical Analysis 3: Comparison: Cohort 3-POSIMIR vs Cohort 3-Placebo; Test type: Superiority; p = 0.1483, ANCOVA; with pooled site and treatment group as factors and incision length as a covariate; LS Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.80 to 0.12], Standard Error of Mean 0.233

2. Primary Outcome: Supplemental Opioid Use
Description: Total morphine-equivalent dose during 0-72 hours post dose. Median values were presented because data was not normally distributed.
Time Frame: 0-72 hours post dose
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Milligram equivalents
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
Milligram equivalents | 87.0 [30.0 to 157.0] | 63.0 [34.0 to 152.0] | 17.0 [8.0 to 26.0] | 22.5 [12.5 to 34.5] | 52.0 [24.0 to 86.6] | 62.0 [24.0 to 86.0]
Statistical Analysis 1: Comparison: Cohort 1-POSIMIR vs Cohort 1-Bupivacaine HCl; Test type: Superiority; p = 0.9901, Wilcoxon (Mann-Whitney); Median Difference (Hodge-Lehmann) = -1.0, 95% CI 2-sided [-54.5 to 52.0]
Statistical Analysis 2: Comparison: Cohort 2-POSIMIR vs Cohort 2-Bupivacaine HCl; Test type: Superiority; p = 0.2010, Wilcoxon Rank-Sum; Median Difference (Hodge-Lehmann) = -5.0, 95% CI 2-sided [-14.0 to 3.4]
Statistical Analysis 3: Comparison: Cohort 3-POSIMIR vs Cohort 3-Placebo; Test type: Superiority; p = 0.5897, Wilcoxon Rank-Sum; Median Difference (Hodge-Lehmann) = -3.0, 95% CI 2-sided [-15.0 to 8.0]

3. Secondary Outcome: Mean Pain Intensity on Movement
Description: Mean pain intensity on movement AUC (time-normalized AUC) during the period 0 to 48 hours post-dose. Pain intensity was assessed with a standard 0 to 10 numeric rating scale (NRS), where no pain at all was rated as 0 and the worst pain imaginable was rated as 10. The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 0 to 48 hours post-dose
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
score on a scale | 5.2 [4.4 to 6.1] | 6.0 [5.0 to 7.0] | 3.2 [2.5 to 4.0] | 4.4 [3.5 to 5.3] | 5.2 [4.8 to 5.5] | 5.5 [5.0 to 5.9]

4. Secondary Outcome: Total Morphine-equivalent Dose
Description: Total morphine-equivalent dose during 0-48 hours post dose.
Time Frame: 0-48 hours post dose
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: mg IV Morphine equivalents
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
mg IV Morphine equivalents | 69.5 [25.0 to 133.0] | 52.0 [29.0 to 122.0] | 15.0 [8.0 to 22.0] | 19.7 [12.5 to 32.5] | 41.5 [21.0 to 66.0] | 43.0 [21.2 to 68.0]

5. Secondary Outcome: Proportion (Percent) of Patients Who Have Evidence of a Wound Infection
Description: From Surgical Wound Healing and Local Tissue Condition Evaluation
Time Frame: 0 to 14 days post-dose (Visits 3 and 4)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
Participants
  Patients with Wound Infection at Visit 3 (Day 7): number analyzed (Participants) | 25 | 15 | 30 | 19 | 122 | 73
  Patients with Wound Infection at Visit 3 (Day 7): yes | 2 | 1 | 0 | 0 | 6 | 0
  Patients with Wound Infection at Visit 3 (Day 7): no | 23 | 14 | 30 | 19 | 116 | 73
  Patients with Wound Infection at Visit 4 (Day 14): number analyzed (Participants) | 24 | 16 | 30 | 19 | 123 | 77
  Patients with Wound Infection at Visit 4 (Day 14): yes | 1 | 2 | 0 | 1 | 4 | 0
  Patients with Wound Infection at Visit 4 (Day 14): no | 23 | 14 | 30 | 18 | 119 | 77

6. Secondary Outcome: Time-to-first Use of Opioid Rescue Medication
Time Frame: 0 to 14 days post-dose (Time from extubation until first opioid use)
Population: ITT Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
Hours | 0.6 [0.2 to 39.2] | 0.5 [0.0 to 6.7] | 0.6 [0.1 to 11.3] | 0.5 [0.1 to 23.9] | 0.6 [0.0 to 22.6] | 0.5 [0.0 to 15.6]

7. Secondary Outcome: Number (Incidence) of Participants With Opioid-related Side Effects
Description: AEs include: nausea, vomiting, constipation, dizziness, somnolence, urinary retention, respiratory depression
Time Frame: 0 to 30 days post-dose
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
Participants | 19 | 10 | 23 | 17 | 93 | 47

8. Secondary Outcome: Pain Intensity at Rest AUC During 0-72 Hours Post Dose
Description: Mean pain intensity at rest AUC during the period 0 to 72 hours post-dose. Pain intensity was assessed with a standard 0 to 10 numeric rating scale (NRS), where no pain at all was rated as 0 and the worst pain imaginable was rated as 10. The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 0-72 hours post dose
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
score on a scale | 3.4 [2.5 to 4.3] | 4.2 [3.2 to 5.2] | 1.7 [1.1 to 2.3] | 2.5 [1.8 to 3.3] | 3.1 [2.7 to 3.5] | 3.5 [3.0 to 3.9]

9. Secondary Outcome: Mean Pain Intensity at Rest AUC During 0-48 Hours Post Dose
Description: Mean pain intensity at rest AUC during the period 0 to 48 hours post-dose. Pain intensity was assessed with a standard 0 to 10 numeric rating scale (NRS), where no pain at all was rated as 0 and the worst pain imaginable was rated as 10. The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 0-48 hours post dose
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
Number analyzed (Participants) | 26 | 17 | 30 | 20 | 126 | 77
score on a scale | 3.6 [2.7 to 4.4] | 4.5 [3.4 to 5.5] | 2.0 [1.4 to 2.6] | 2.9 [2.1 to 3.6] | 3.4 [3.0 to 3.8] | 3.8 [3.4 to 4.3]

ADVERSE EVENTS:
Arm/Group | Cohort 1-POSIMIR | Cohort 1-Bupivacaine HCl | Cohort 2-POSIMIR | Cohort 2-Bupivacaine HCl | Cohort 3-POSIMIR | Cohort 3-Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/18 | 0/30 | 0/20 | 1/129 | 0/78
Serious Adverse Events (participants affected / at risk) | 9/30 | 4/18 | 0/30 | 1/20 | 16/129 | 9/78
Other Adverse Events (participants affected / at risk) | 30/30 | 17/18 | 28/30 | 20/20 | 126/129 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-POSIMIR (N=30) | Cohort 1-Bupivacaine HCl (N=18) | Cohort 2-POSIMIR (N=30) | Cohort 2-Bupivacaine HCl (N=20) | Cohort 3-POSIMIR (N=129) | Cohort 3-Placebo (N=78)
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 6 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Application site discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-POSIMIR (N=30) | Cohort 1-Bupivacaine HCl (N=18) | Cohort 2-POSIMIR (N=30) | Cohort 2-Bupivacaine HCl (N=20) | Cohort 3-POSIMIR (N=129) | Cohort 3-Placebo (N=78)
Nausea (Gastrointestinal disorders) | 16 (18) | 9 (11) | 17 (23) | 14 (20) | 77 (80) | 40 (42)
Vomiting (Gastrointestinal disorders) | 9 (12) | 2 (2) | 9 (13) | 7 (10) | 23 (26) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 8 (8) | 8 (8) | 23 (23) | 8 (8)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6) | 3 (3) | 16 (19) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (3) | 2 (3) | 16 (16) | 10 (10)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 10 (10) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (4) | 0 (0) | 4 (4) | 4 (4)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site discolouration (General disorders) | 14 (17) | 6 (7) | 15 (18) | 4 (5) | 80 (116) | 46 (66)
Pyrexia (General disorders) | 7 (7) | 3 (3) | 2 (2) | 1 (1) | 14 (14) | 11 (11)
Fatigue (General disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 3 (3)
Chest pain (General disorders) | 3 (3) | 0 (0) | 3 (6) | 1 (6) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 | 2 (2) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 11 (15) | 1 (1) | 9 (9) | 12 (12)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 7 (7) | 4 (5) | 13 (13) | 6 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 18 (18) | 3 (3)
Wound secretion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 14 (15) | 6 (7)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 4 (4)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 9 (10) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 8 (8)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10) | 2 (2) | 0 (0) | 0 (0) | 14 (14) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (8) | 5 (5) | 9 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 8 (18) | 7 (9) | 6 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 8 (8) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 10 (11) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 8 (8) | 7 (7)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 13 (13) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 2 (2)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes